CLINICAL TRIAL: NCT05204264
Title: A Randomized Single-blind Trial in Adult Population With Anxiety Disorders: Comparison of a Mindfulness-based Emotional Regulation Program Versus an Acceptance and Commitment Therapy-based Intervention
Brief Title: Mindfulness-based Emotional Regulation Versus ACT in Anxiety
Acronym: MER-ACT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, Dr. Eduardo Fernández-Jiménez, Principal Investigator, Hospital Universitario La Paz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5373
Record Dates: First submitted 2022-01-11; First posted 2022-01-24 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: Anxiety
Keywords: Acceptance and Commitment Therapy; Mindfulness-based Emotional Regulation; Randomized clinical trial; Neuropsychology
MeSH Terms: conditions — Anxiety Disorders | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be randomized according to the score on the Acceptance and Action Questionnaire-II (blocking factor) without knowing the treatment they were allocated to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acceptance and Commitment Therapy (ACT) (Experimental): Intervention based on Acceptance and Commitment Therapy that promotes the acceptance and defusion of unwanted internal experiences and commitment to values of the personal life project.
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT)
- Mindfulness-based Emotional Regulation (MER) (Experimental): Intervention inspired in the Mindfulness-Based Stress Reduction program that fosters the development of a behavioral pattern made up of conscious responses in order to decrease reactivity to stressors.
  Interventions: Behavioral: Mindfulness-based Emotional Regulation (MER)

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy (ACT) — This intervention uses techniques based on mindfulness, metaphors and exposition exercises both in imagination and in real contexts.
  Arms: Acceptance and Commitment Therapy (ACT)
Behavioral: Mindfulness-based Emotional Regulation (MER) — This intervention includes both formal practices of body scan meditation, standing / sitting Hatha yoga, meditations focused on the breath or other objects of attention, exercises of benevolence or kindness with affection (loving-kindness); as well as informal mindfulness practices in activities of daily living.
  Arms: Mindfulness-based Emotional Regulation (MER)

SUMMARY:
Background: There is a paucity of randomized clinical trials which address the relationship between training in mindfulness and neuropsychological outcomes. Also, how psychotherapeutic interventions were delivered before and during the COVID-19 pandemic and its possible differential results need more scientific attention.

Aims: To compare the effectiveness of an intervention based on the Acceptance and Commitment Therapy (ACT) versus a Mindfulness-based Emotional Regulation (MER) intervention among adult patients with anxiety disorders.

Methods: This randomized, single-blind, clinical trial is being conducted in a community Mental Health Unit (Colmenar Viejo, Madrid) in Spain. Potential outpatients will be over 18 years (until 75 years) with some type of specific or unspecified anxiety disorder. They will be assessed for inclusion/exclusion criteria and randomized according to the score on the Acceptance and Action Questionnaire-II (used as a blocking factor). One of the interventions was adapted from the Acceptance and Commitment Therapy (ACT) for anxiety disorders and MER was based on the Mindfulness-Based Stress Reduction program. Each intervention has been designed to be weekly, during 8 weeks, guided by two Clinical Psychology residents. Interventions have been delivered face-to-face before the COVID-19 pandemic, or via online currently. A 2x3 mixed-factorial ANOVA (intervention type x pre-treatment, post-treatment and 6-month follow-up) will be conducted, with Sidak-correction post hoc tests. The primary measures are the TMT score (A and B forms), Stroop test, Digit span subtests from the Wechsler Adult Intelligence Scale, version IV (Forward, Backward and Sequencing subtests), Acceptance and Action Questionnaire-II, and Anxiety Sensitivity Index-3 (ASI-3). Secondary measures are the Five Facets Mindfulness Questionnaire (FFMQ), Toronto Alexithymia Scale 20-item (TAS-20), Reflective Functioning Questionnaire (RFQ-8), Hospital Anxiety and Depression Scale (HADS), and the World Health Organization's Quality of Life Questionnaire (WHOQOL-BREF). Norms based on the Spanish general population will be used.

Results: This clinical trial started in February 2019 and it is expected to end in September 2023. The minimum sample size required is 128 participants (64 each intervention) to achieve medium effect sizes on primary outcomes (alfa = .05 and beta = .20). So far, 107 adult patients with anxiety disorders participated (64 participants in face-to-face interventions before the COVID-19 pandemic; and 43 participants via online, during the pandemic).

Conclusions: This is the first study to compare two mindfulness-based interventions on several neurocognitive functions and other psychological domains among adult patients with anxiety disorders.

ELIGIBILITY:
Inclusion Criteria:

* Spanish as mother tongue or a very high level in Spanish to understand the patient information sheet, the informed consent, as well as being able to follow the group intervention sessions and the homework.
* Diagnosis of an anxiety disorder, avoidant personality disorder, adjustment disorders with anxious/anxious-depressive symptomatology, as well as unspecified anxiety disorders.

Exclusion Criteria:

* Continuing individual psychotherapeutic treatment from the beginning of the group intervention until the end of it.
* Other diagnoses of severe mental disorder; cluster A or B personality disorders; and/or substance use disorder in the past 6 months.
* Diagnosis of intellectual disability, mild cognitive impairment or dementia.
* Changes in psychopharmacological treatment (in active ingredient or doses) in the month before each intervention.
* Diagnosis of uncontrolled or non-stabilized organic disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2019-02-18 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Trail Making Test (TMT) | Baseline
  It evaluates selective/alternative visual attention by the time of execution (seconds)
Trail Making Test (TMT) | 2 months
  It evaluates selective/alternative visual attention by the time of execution (seconds)
Trail Making Test (TMT) | 8 months
  It evaluates selective/alternative visual attention by the time of execution (seconds)
Stroop Color-Word Interference Test | Baseline
  It measures processing speed and visual inhibitory control by the total number of items achieved
Stroop Color-Word Interference Test | 2 months
  It measures processing speed and visual inhibitory control by the total number of items achieved
Stroop Color-Word Interference Test | 8 months
  It measures processing speed and visual inhibitory control by the total number of items achieved
Digit span subtests from the Wechsler Adult Intelligence Scale, version IV (WAIS-IV): Forward, Backward and Sequencing subtests | Baseline
  It evaluates span of immediate recall and verbal working memory by the total number of items achieved and the maximum number of remembered elements
Digit span subtests from the Wechsler Adult Intelligence Scale, version IV (WAIS-IV): Forward, Backward and Sequencing subtests | 2 months
  It evaluates span of immediate recall and verbal working memory by the total number of items achieved and the maximum number of remembered elements
Digit span subtests from the Wechsler Adult Intelligence Scale, version IV (WAIS-IV): Forward, Backward and Sequencing subtests | 8 months
  It evaluates span of immediate recall and verbal working memory by the total number of items achieved and the maximum number of remembered elements
The Acceptance and Action Questionnaire-II (AAQ-II) | Baseline
  It evaluates experiential avoidance and psychological inflexibility. It is a 7-item self-report instrument, rated on a 7-point Likert scale, with a total scale score ranging from 7 to 49. Higher scores indicate higher levels of experiential avoidance and psychological inflexibility
The Acceptance and Action Questionnaire-II (AAQ-II) | 2 months
  It evaluates experiential avoidance and psychological inflexibility. It is a 7-item self-report instrument, rated on a 7-point Likert scale, with a total scale score ranging from 7 to 49. Higher scores indicate higher levels of experiential avoidance and psychological inflexibility
The Acceptance and Action Questionnaire-II (AAQ-II) | 8 months
  It evaluates experiential avoidance and psychological inflexibility. It is a 7-item self-report instrument, rated on a 7-point Likert scale, with a total scale score ranging from 7 to 49. Higher scores indicate higher levels of experiential avoidance and psychological inflexibility
The Anxiety Sensitivity Index-3 (ASI-3) | Baseline
  It measures concerns associated with possible negative consequences of anxiety-related symptoms in three dimensions (physical, cognitive and social). It is an 18-item self-report, rated on a 5-point Likert scale, with a total scale score (ranging from 0 to 72) and three 6-item subscales (Physical, Cognitive and Social Concerns, ranging from 0 to 24 points each). Higher scores indicate higher anxiety sensitivity
The Anxiety Sensitivity Index-3 (ASI-3) | 2 months
  It measures concerns associated with possible negative consequences of anxiety-related symptoms in three dimensions (physical, cognitive and social). It is an 18-item self-report, rated on a 5-point Likert scale, with a total scale score (ranging from 0 to 72) and three 6-item subscales (Physical, Cognitive and Social Concerns, ranging from 0 to 24 points each). Higher scores indicate higher anxiety sensitivity
The Anxiety Sensitivity Index-3 (ASI-3) | 8 months
  It measures concerns associated with possible negative consequences of anxiety-related symptoms in three dimensions (physical, cognitive and social). It is an 18-item self-report, rated on a 5-point Likert scale, with a total scale score (ranging from 0 to 72) and three 6-item subscales (Physical, Cognitive and Social Concerns, ranging from 0 to 24 points each). Higher scores indicate higher anxiety sensitivity

SECONDARY OUTCOMES:
The Five Facets of Mindfulness Questionnaire (FFMQ) | Baseline
  It is a self-report instrument of 39 items, rated on a 5-point Likert scale, that are grouped into both a total scale score (with a mean score ranging from 1 to 5) and five specific subscales: Observing (8 items), Describing (8 items), Acting with awareness (8 items), Non-judgment (8 items), and Non-reactivity (7 items). Higher values indicate higher levels in each domain
The Five Facets of Mindfulness Questionnaire (FFMQ) | 2 months
  It is a self-report instrument of 39 items, rated on a 5-point Likert scale, that are grouped into both a total scale score (with a mean score ranging from 1 to 5) and five specific subscales: Observing (8 items), Describing (8 items), Acting with awareness (8 items), Non-judgment (8 items), and Non-reactivity (7 items). Higher values indicate higher levels in each domain
The Five Facets of Mindfulness Questionnaire (FFMQ) | 8 months
  It is a self-report instrument of 39 items, rated on a 5-point Likert scale, that are grouped into both a total scale score (with a mean score ranging from 1 to 5) and five specific subscales: Observing (8 items), Describing (8 items), Acting with awareness (8 items), Non-judgment (8 items), and Non-reactivity (7 items). Higher values indicate higher levels in each domain
The Toronto Alexithymia Scale 20-item (TAS-20) | Baseline
  It is a self-report instrument that measures both a global factor of alexithymia, and three specific domains: Difficulty in Identifying Feelings (7 items), Difficulty in Describing Feelings (5 items) and Externally Oriented Thinking (8 items). Items are rated on a 5-point Likert scale. The total scale score ranges between 20 and 100, with higher scores indicating greater level of alexithymia
The Toronto Alexithymia Scale 20-item (TAS-20) | 2 months
  It is a self-report instrument that measures both a global factor of alexithymia, and three specific domains: Difficulty in Identifying Feelings (7 items), Difficulty in Describing Feelings (5 items) and Externally Oriented Thinking (8 items). Items are rated on a 5-point Likert scale. The total scale score ranges between 20 and 100, with higher scores indicating greater level of alexithymia
The Toronto Alexithymia Scale 20-item (TAS-20) | 8 months
  It is a self-report instrument that measures both a global factor of alexithymia, and three specific domains: Difficulty in Identifying Feelings (7 items), Difficulty in Describing Feelings (5 items) and Externally Oriented Thinking (8 items). Items are rated on a 5-point Likert scale. The total scale score ranges between 20 and 100, with higher scores indicating greater level of alexithymia
The Reflective Functioning Questionnaire (RFQ-8) | Baseline
  It is an 8-item self-report instrument, rated on a 7-point Likert scale, that assesses the degree of certainty or uncertainty about their own or someone else's mental states. It includes two subscales (with a double-scoring procedure): Uncertainty about mental states (5 items, with range 0-3) and Certainty about mental states (6 items, with range 0-2). High levels of certainty about mental states indicate hypermentalizing and high levels of uncertainty indicate hypomentalizing
The Reflective Functioning Questionnaire (RFQ-8) | 2 months
  It is an 8-item self-report instrument, rated on a 7-point Likert scale, that assesses the degree of certainty or uncertainty about their own or someone else's mental states. It includes two subscales (with a double-scoring procedure): Uncertainty about mental states (5 items, with range 0-3) and Certainty about mental states (6 items, with range 0-2). High levels of certainty about mental states indicate hypermentalizing and high levels of uncertainty indicate hypomentalizing
The Reflective Functioning Questionnaire (RFQ-8) | 8 months
  It is an 8-item self-report instrument, rated on a 7-point Likert scale, that assesses the degree of certainty or uncertainty about their own or someone else's mental states. It includes two subscales (with a double-scoring procedure): Uncertainty about mental states (5 items, with range 0-3) and Certainty about mental states (6 items, with range 0-2). High levels of certainty about mental states indicate hypermentalizing and high levels of uncertainty indicate hypomentalizing
The Hospital Anxiety and Depression Scale (HADS) | Baseline
  It measures anxious and depressive symptomatology. It is a 14-item self-report, rated on a 4-point Likert scale, with a total score (ranging from 0 to 42) and two subscales (7 items each, ranging from 0-21)
The Hospital Anxiety and Depression Scale (HADS) | 2 months
  It measures anxious and depressive symptomatology. It is a 14-item self-report, rated on a 4-point Likert scale, with a total score (ranging from 0 to 42) and two subscales (7 items each, ranging from 0-21)
The Hospital Anxiety and Depression Scale (HADS) | 8 months
  It measures anxious and depressive symptomatology. It is a 14-item self-report, rated on a 4-point Likert scale, with a total score (ranging from 0 to 42) and two subscales (7 items each, ranging from 0-21)
The World Health Organization's Quality of Life Questionnaire (WHOQOL-BREF) | Baseline
  It is a self-report instrument of 26 items grouped into general health questions (2 items) and four factors: Physical Health (7 items), Psychological Health (6 items), Social Relations (3 items) and Environment (8 items), ranging from 0 to 100 points. Higher scores in each domain indicate higher level of satisfaction
The World Health Organization's Quality of Life Questionnaire (WHOQOL-BREF) | 2 months
  It is a self-report instrument of 26 items grouped into general health questions (2 items) and four factors: Physical Health (7 items), Psychological Health (6 items), Social Relations (3 items) and Environment (8 items), ranging from 0 to 100 points. Higher scores in each domain indicate higher level of satisfaction
The World Health Organization's Quality of Life Questionnaire (WHOQOL-BREF) | 8 months
  It is a self-report instrument of 26 items grouped into general health questions (2 items) and four factors: Physical Health (7 items), Psychological Health (6 items), Social Relations (3 items) and Environment (8 items), ranging from 0 to 100 points. Higher scores in each domain indicate higher level of satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Fernández-Jiménez, PhD, Principal Investigator — Hospital Universitario La Paz
Locations (1):
- Centro de Salud Mental de Colmenar Viejo Sur, Colmenar Viejo, Madrid, Spain

REFERENCES:
- See also: Attentional functioning after two online mindfulness-based group interventions: Acceptance and commitment therapy and a mindfulness-based emotional regulation intervention in anxiety disorders. Preliminary results. — https://www.cambridge.org/core/journals/european-psychiatry/article/attentional-functioning-after-two-online-mindfulnessbased-group-interventions-acceptance-and-commitment-therapy-and-a-mindfulnessbased-emotional-regulation-intervention-in-anxiety-disorders-preliminary-results/27B4F47CF42CC21F6310B1134E1B6F03
- See also: On gender and cognitive flexibility. The REM-ACT study: Acceptance and commitment therapy versus a mindfulness-based emotional regulation intervention in anxiety disorders. A randomized controlled trial. — https://www.cambridge.org/core/journals/european-psychiatry/article/on-gender-and-cognitive-flexibility-the-remact-study-acceptance-and-commitment-therapy-versus-a-mindfulnessbased-emotional-regulation-intervention-in-anxiety-disorders-a-randomized-controlled-trial/F3FB2263F89DECFA3F098155EB15553B
- See also: On gender and stroop effect. The REM-ACT study: Acceptance and commitment therapy versus a mindfulness-based emotional regulation intervention in anxiety disorders. A randomized controlled trial. — https://www.cambridge.org/core/journals/european-psychiatry/article/on-gender-and-stroop-effect-the-remact-study-acceptance-and-commitment-therapy-versus-a-mindfulnessbased-emotional-regulation-intervention-in-anxiety-disorders-a-randomized-controlled-trial/7E2CE606A976E7B199F0447183AF092D
- See also: TMT-B after two online mindfulness-based group interventions: Acceptance and commitment therapy and a mindfulness-based emotional regulation intervention in anxiety disorders. Preliminary results. — https://www.cambridge.org/core/journals/european-psychiatry/article/tmtb-after-two-online-mindfulnessbased-group-interventions-acceptance-and-commitment-therapy-and-a-mindfulnessbased-emotional-regulation-intervention-in-anxiety-disorders-preliminary-results/3687B32F066BD1751CE336437B3B9739
- See also: On gender and TMT-A. The REM-ACT study: Acceptance and commitment therapy versus a mindfulness-based emotional regulation intervention in anxiety disorders. A randomized controlled trial. — https://www.cambridge.org/core/journals/european-psychiatry/article/on-gender-and-tmta-the-remact-study-acceptance-and-commitment-therapy-versus-a-mindfulnessbased-emotional-regulation-intervention-in-anxiety-disorders-a-randomized-controlled-trial/0B7FED243C851DB16EAAB1EC22569EED